CLINICAL TRIAL: NCT03024229
Title: The Importance of Metabolomics in Assessing the Quality of Kidney Transplants Retained on a LifePort® Perfusion Machine Before Renal Transplantation
Brief Title: Metabolomics in Assessing the Quality of Kidney Transplants Retained on a LifePort® Perfusion Machine
Acronym: RENALIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Laboratory of Biochemistry, University François Rabelais of TOURS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PHAO15/FB-RENALIFE
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Renal Transplantation
Keywords: Transplantation;perfusion machine

STUDY DESIGN:
Intervention Model Description: Metabolic assessment in Urine and perfusion liquids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LifePort® perfusion machine (Other): Metabolomic analysis of the preservation fluid of the graft, donor and recipient urine by nuclear magnetic resonance spectroscopy, and if possible by liquid and gas chromatography coupled with mass spectrometry.
  Interventions: Device: LifePort® perfusion machine

INTERVENTIONS:
Device: LifePort® perfusion machine — Renal perfusion on LifePort® machine

SUMMARY:
When the kidneys are perfused on perfusion machines before transplantation, the resistance parameters as well as the histological score on the pre-implantation biopsy participate in the evaluation of the quality of the graft. The metabolomic profile of the infusion fluid could provide additional evidence.

DETAILED DESCRIPTION:
The quality of the renal transplant prior to transplantation is essential for the recovery of graft function in the days following transplantation and its long-term survival. When the kidneys are perfused on perfusion machines before transplantation, the resistance parameters as well as the histological score on the pre-implantation biopsy participate in the evaluation of the quality of the graft. The metabolomic profile of the infusion fluid could provide additional evidence.

ELIGIBILITY:
Inclusion Criteria:

* Donors aged 18 years or more in brain death or who died of cardiac arrest collected locally in Tours, associated with the major local recipients of the grafts over the same period.

Exclusion Criteria:

* Kidney transplant removed but stored in a static preservative.
* Kidney grafts of donors aged 18 years or more, removed and not retained on a LifePort® perfusion machine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
IGF | 7 days
  Immediate Graft Function (IGF), defined by serum creatinine less than 250 μM / L at day 7 post-kidney transplant, without requiring dialysis of the recipient patient.

SECONDARY OUTCOMES:
DGF | 7 days
  DGF Delayed graft function : Dialysis need within 7 days post-transplant
BANFF-1 | PRE-OPERATIONAL
  Anatomo-pathological classification of the pre-implantation biopsy according to the revised Banff classification 2013
BANFF-2 | 3 months
  Anatomo-pathological classification of systematic biopsy at 3 months post-transplant according to the revised Banff classification 2013

CONTACTS AND LOCATIONS:
Overall Officials: Franck BRUYERE, MD-PhD, Principal Investigator — University François Rabelais of TOURS
Locations (2):
- France (2):
  - Urology CHRU-TOURS, Tours, I&L
  - CHR-ORLEANS Service d'Urologie, Orléans, Loiret

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Faucher Q, Alarcan H, Sauvage FL, Forestier L, Miquelestorena-Standley E, Nadal-Desbarats L, Arnion H, Venhard JC, Brichart N, Bruyere F, Marquet P, Barin-Le Guellec C. Perfusate Metabolomics Content and Expression of Tubular Transporters During Human Kidney Graft Preservation by Hypothermic Machine Perfusion. Transplantation. 2022 Sep 1;106(9):1831-1843. doi: 10.1097/TP.0000000000004129. Epub 2022 Apr 20. PMID 35442245